CLINICAL TRIAL: NCT07050264
Title: The Effect of Simulated Burn Injury on Post Exercise Recovery in Hot Environments
Acronym: HSR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine and director of the thermal and vascular physiology lab, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU20251344; R35GM152112-01 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Burn Injury; Body Temperature Regulation; Cardiovascular Physiology
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hot and Humid with simulated burns (Experimental): Individuals will be exposed to hot and humid conditions with a simulated burn injury.
  Interventions: Other: Simulated burn injury via application of absorbent and impermeable material over 60% of the body
- Hot and Humid without simulated burns (No Intervention): Individuals will be exposed to hot and humid conditions without a simulated burn injury.
- Hot and Dry with simulated burns (Experimental): Individuals will be exposed to hot and dry conditions with a simulated burn injury.
  Interventions: Other: Simulated burn injury via application of absorbent and impermeable material over 60% of the body
- Hot and Dry without simulated burns (No Intervention): Individuals will be exposed to hot and dry conditions without a simulated burn injury.

INTERVENTIONS:
Other: Simulated burn injury via application of absorbent and impermeable material over 60% of the body — Simulated burn injury via application of absorbent and impermeable material over 60% of the body
  Arms: Hot and Dry with simulated burns; Hot and Humid with simulated burns

SUMMARY:
Burn survivors have difficulty thermoregulating due to reduced skin blood flow and sweating responses at the grafted sites. It has been previously shown that this impaired heat dissipation results in burn survivors experiencing higher core temperatures for a given exercise/environmental exposure compared to non-burned individuals. This also holds true with the use of simulated burn injury. When an absorbent material is applied to the skin over a desired amount of body surface area, it replicates a burn injury of the same size (i.e., simulated burn injury). A question that remains unknown is if this impaired thermoregulation in burn survivors would affect post-exercise core temperature recovery, i.e., do burn survivors recover slower than non-burned individuals upon stopping exercise. To that end, the primary objective of this project is to determine the rate at which body temperature and other markers of thermoregulation recover after a bout of exercise in the heat and if this response is different in the same individual with and without simulated burn injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years of age
* free of any significant underlying medical problems based upon a detailed medical history and physical exam, and normal resting electrocardiogram.

Exclusion Criteria:

* Known heart disease
* other chronic medical conditions requiring regular medical therapy including cancer, diabetes, neurological diseases, and uncontrolled hypertension, etc. as well as serious abnormalities detected on routine screening.
* Individuals who are pregnant, planning to become pregnant, or breastfeeding will be excluded, this will be confirmed in females using a urine pregnancy test.
* Taking prescribed medications (such as beta blockers and non-dihydropyridine calcium channel blockers) or over-the-counter medications that have known influences on thermoregulatory response.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* body mass index is ≥ 31 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Core Temperature | From baseline to end of 60 minutes of recovery

SECONDARY OUTCOMES:
Heart Rate | From baseline to the end of 60 minutes of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Craig G Crandall, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine - Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No